CLINICAL TRIAL: NCT03688191
Title: Sirolimus in Patients With Connective Tissue Disease Related Thrombocytopenia (CTD-TP): a Single-arm, Open-label Clinical Trial in China
Brief Title: Study of Sirolimus in CTD-TP in China
Acronym: SSCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SirolimusforCTD-IP
Record Dates: First submitted 2018-07-30; First posted 2018-09-28 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2018-12

CONDITIONS: Connective Tissue Diseases; Thrombocytopenia
Keywords: Sirolimus; connective tissue disease; thrombocytopenia
MeSH Terms: conditions — Connective Tissue Diseases; Thrombocytopenia | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): participants who received sirolimus treatment
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Patients will receive oral sirolimus at a starting dose of 2 mg per day for 3 days and a sequential dose of 1mg per day, with dose adjusted according to tolerance and to maintain a therapeutic range of 6-15 ng/mL.

SUMMARY:
We have designed a single-arm, open-label study of sirolimus in Chinese patients with refractory CTD-TP unresponsive to, or intolerant of, conventional medications at Peking Union Medical College Hospital (PUMCH). Patients received oral sirolimus at a starting dose of 2 mg per day for 3 days and a sequential dose of 1mg per day, with dose adjusted according to tolerance and to maintain a therapeutic range of 6-15 ng/mL. Patients were treated with sirolimus for more than 6 months. Safety outcomes and the efficacy endpoints were assessed in all patients who received at least one dose of treatment.

DETAILED DESCRIPTION:
Connective tissue disease related thrombocytopenia (CTD-TP) is one of the common visceral complications of connective tissue diseases (CTD) with a poor response to traditional therapy. To date, some successful cases were reported in sirolimus treating refractory CTD-TP as a newly therapeutic method. However, there is still a lack of prospective clinical trials. This study aims to evaluate the efficacy of sirolimus in the treatment of refractory CTD-TP. To investigate this issue, investigators have designed a single-arm, open-label clinical trial of refractory CTD-TP patients in Peking Union Medical College Hospital (PUMCH). In this study, the researchers will enroll 20 patients who have a poor response to at least 6 months' traditional treatment. The participants will receive oral sirolimus treatment for 12 months. The primary end point is the change of platelet count in CBC. Secondary end points include the change of CTD activity, the time to disease complete remission and all-cause serious adverse events (SAE).

Research Question:

Does sirolimus improve the prognosis in patients with connective tissue disease related thrombocytopenia (CTD-TP) in Chinese patients?

Specific aims:

1. To determine the efficacy of sirolimus for the treatment of CTD-TP in Chinese patients
2. To evaluate the safety of sirolimus for the treatment of CTD-TP in Chinese patients
3. To analyze the clinical characteristics of CTD-TP in the sirolimus effective patients

Methods:

This is a prospective open-label trial in a period of 12 months. Thrombocytopenia is defined that the count of platelet is less than 100×109/L. CTDs include SLE, pSS, RA, scleroderma, RA, dermatomyositis and MCTD. The newly diagnosed CTD-TP patients who have received no steroid or IS treatment will be ruled out the trial. All the participants should fulfill one of the criteria of SLE, pSS, RA, scleroderma, RA, dermatomyositis and MCTD and suffer from refractory TP, or be diagnosed CTD-associated TP by two experimental rheumatologists. The current standard treatment for CTD-TP is glucocorticoid plus one kind of immunosuppressant. The patients who still have TP after more than 3 months' standard treatment will be included into the trial. After signing informed consent forms, participants will receive oral sirolimus at a starting dose of 2 mg per day for 3 days and a sequential dose of 1mg per day, with dose adjusted according to tolerance and to maintain a therapeutic range of 6-15 ng/mL. Baseline data will be collected at enrollment. All participants will finish their 5 follow-up assessments (1st mon, 2nd mon, 4th mon, 6th mon and 12th mon) in 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory CTD-TP unresponsive to, or intolerant of, conventional medications at Peking Union Medical College Hospital.

Exclusion Criteria:

* new diagnosed CTD-IT patients

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with complete remission of platelet count | 6 months
  Complete remission of platelet count means the platelet count over 100X10^9/L. every participants will take CBC as their screening times.

SECONDARY OUTCOMES:
Number of participants with partial remission of platelet count | 6 months
  Partial remission of ITP means that the platelet count was less than 100X10^9/L, but it was more than two times higher than that before treatment.

OTHER OUTCOMES:
Bleeding Events with treatment-related adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Peng, Professor, Study Chair — Peking Union Medical College Hospital; Chanyuan WU, MD, Principal Investigator — Peking Union Medical College Hospital; Mengtao LI, Professor, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Study of Sirolimus in CTD-IP in China

REFERENCES:
- [Derived] Wu C, Wang Q, Xu D, Li M, Zeng X. Sirolimus for patients with connective tissue disease-related refractory thrombocytopenia: a single-arm, open-label clinical trial. Rheumatology (Oxford). 2021 Jun 18;60(6):2629-2634. doi: 10.1093/rheumatology/keaa645. PMID 33200217